CLINICAL TRIAL: NCT05155020
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of AK120 in the Treatment of Subjects With Moderate-to-severe Asthma
Brief Title: A Study to Evaluate the Efficacy and Safety of AK120 in the Treatment of Subjects With Moderate-to-severe Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The clinical development strategy has been changed
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK120-201
Record Dates: First submitted 2021-12-01; First posted 2021-12-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Asthma
Keywords: AK120; Efficacy; Safety
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AK120 regimen 1 (Experimental)
  Interventions: Biological: AK120
- AK120 regimen 2 (Experimental)
  Interventions: Biological: AK120
- AK120 regimen 3 (Experimental)
  Interventions: Biological: AK120
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AK120 — AK120 regimen 1-subcutaneous injection every two weeks up to week 24, and follow up to week 32.
  Arms: AK120 regimen 1
Biological: AK120 — AK120 regimen 2(first dose doubling)-subcutaneous injection and then every two weeks up to week 24, and follow up to week 32.
  Arms: AK120 regimen 2
Biological: AK120 — AK120 regimen 3(first dose doubling)-subcutaneous injection and then every two weeks up to week 24, and follow up to week 32.
  Arms: AK120 regimen 3
Biological: Placebo — Placebo subcutaneous injection every two weeks up to week 24, and follow up to week 32.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, phase II clinical study to evaluate the efficacy and safety of AK120 in the treatment of subjects with moderate-to-severe asthma.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter, phase II clinical study. The purpose of this study is to evaluate the efficacy and safety of AK120 in the treatment of subjects with moderate-to-severe asthma and not adequately controlled with current stable medium-to-high-dose inhaled glucocorticoids plus up to two additional controllers.Subjects will be randomized to receive AK120 or placebo subcutaneous injection.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subjects aged ≥18 years old and ≤75 years old;
2. Asthma was diagnosed ≥ 12 months before screening, current stable treatment with medium-to-high-dose inhaled glucocorticoids plus up to two additional controllers ≥ 3 months;
3. Blood eosinophil≥ 200 cells per microliter within 6 months before screening;
4. During the screening, 40% of the predicted normal value < pre-bronchodilator FEV1 < 80% of the predicted normal value, within 12 months before randomization, reversible airflow restriction was recorded;
5. Asthma was inadequately controlled;
6. For women with childbearing potential, they are not pregnant or lactating, and the subjects and their partners voluntarily take effective contraceptive measures judged by the investigators during the treatment and at least 3 months after last dose.

Key Exclusion Criteria:

1. Subjects with lung diseases other than asthma, which may affect the subject's health or end point evaluation of the study;
2. Subjects had severe exacerbation events or systemic glucocorticoids usage within 1 month before randomization;
3. Respiratory tract infection and any serious infection within 1 month before randomization;
4. Subjects with parasitic infection, active tuberculosis infection, Hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or syphilis positive confirmation test;
5. Known or suspected history of immunosuppression;
6. History of malignant tumors;
7. A history of smoking: those who had quit smoking for ≤ 6 months before screening, or smoking history > 10 pack per year;
8. Previous treatment with interleukin-4 (IL-4) or interleukin-13 (IL-13) inhibitors, and inadequate washout period of other biologic therapy;
9. Allergen immunotherapy within 3 months before randomization;
10. Progressive or uncontrolled other diseases or any other conditions or abnormal laboratory tests for which the investigator assess that the subjects are not suitable to enrol in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Change in pre-bronchodilator forced expiratory volume in 1 second (FEV1) from baseline at week 12. | At week 12

SECONDARY OUTCOMES:
Annualized rate of severe exacerbation events within 24 weeks. | Baseline to Week24
Annualized rate of severe exacerbation events within 32 weeks. | Baseline to Week32
Change in pre-bronchodilator FEV1 from baseline to week 32. | Baseline to Week32
Percentage change in pre-bronchodilator FEV1 from baseline to week 32. | Baseline to Week32
Change in post-bronchodilator FEV1 from baseline to week 32. | Baseline to Week32
Change in fractional exhaled nitric oxide (FeNO) from baseline to week 32. | Baseline to Week32
Changes in asthma control questionnaire (ACQ-5) scores from baseline to week 32. | Baseline to Week32
Change in standardized version of the asthma quality of life (AQLQ-s) scores from baseline at week 12 and 24. | at week 12,week 24
Safety assessment: treatment-emergent adverse events (TEAE), serious adverse events (SAE) . | Baseline to Week32
Pharmacokinetics (PK): AK120 concentration at different time points. | Baseline to Week32
Immunogenicity assessment: number and percentage of subjects with detectable anti-AK120 antibody (ADA). | Baseline to Week32

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Jingmei General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Luoyang Central Hospital, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Baogang Hospital, Inner Mongolia, China, Baotou, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangxi Provincial Prople's Hospita, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated Hospital Zhejiang University School of Medicine,, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No